CLINICAL TRIAL: NCT06578494
Title: The Efficacy of Implementing Nurse-performed Ultrasound-guided Peripheral Intravenous Access in Oncology Patients: a Prospective Interventional Clinical Study
Brief Title: The Efficacy of Implementing Nurse-performed Ultrasound-guided Peripheral Intravenous Access in Oncology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faroese Hospital System (Other)
Collaborators: National Hospital of the Faroe Islands (Other Government); University of the Faroe Islands (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ultrasound IV
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Supportive Care
Keywords: Ultrasonography; Intravenous; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: This is a before and after study, where the patients pre-implementation stage receive intravenous access via the traditional palpation technique and in the post-implementation stage receive ultrsound-guided intravenous cannulation.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided peripheral intravenous access (Experimental): The patients in the experimental arm will receive ultrasound-guided peripheral intravenous catheter placement, where the dynamic needle tip (DNTP) approach (short-axis) will be used.
  Interventions: Device: Ultrasound
- Traditional palpation intravenous access technique (Active Comparator): The comparator group will receive the traditional palpation intravenous access technique.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound-guided peripheral intravenous catheter insertion

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of nurse-performed ultrasound-guided intravenous access in oncology patients on the oncological outpatient unit in the National Hospital of the Faroe Islands.

DETAILED DESCRIPTION:
This project is prospective, interventional, clinical study aligned in four different time stages.

In the first stage, the pre-implementation stage, procedures are as usual, where the patient receives intravenous access via the use of the traditional palpation technique and data will be registered. In the next stage, the training stage, the nurses on the oncological outpatient unit will be trained in the use of the ultrasound-guided technique to place peripheral intravenous catheters and will be supervised by specialists in ultrasound. In the third stage, the implementation stage, the nurses will use the ultrasound technique as a daily routine in their practice. In the fourth stage, the post-implementation stage, the same data registration as in the first stage will be registered (see outcome measures) and the results will be compared in order to see the efficacy before and after implementation of ultrasound guidance. It is estimated a total sample of 100 cannulation procedures with approximately 30 patients needed in the pre-implementation and post-implementation stages.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients admitted to the oncological outpatient unit are eligible for inclusion if they are scheduled for treatment with chemotherapy requiring placement of peripheral intravenous catheter, aged 18 years or older, and reside in the Faroe Islands.

Exclusion Criteria:

* Lack of informed consent and mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2025-10-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate | The time frame for the outcome measure first attempt succes rate for each participant is estimated 1 hour in the pre-implementation stage and 1 hour in the post-implementation stage.
  Placement of a functional peripheral intravenous catheter on the first attempt. Defined as retraction of the needle, blood in the plastic catheter, smooth insertion of the plastic catheter and subsequent flush with isotonic saline without signs of extravasal placement.

SECONDARY OUTCOMES:
Number of skin punctures | The time frame for the outcome measure number of attempts for each participant is estimated 1 hour in the pre-implementation stage and 1 hour in the post-implementation stage.
  Total number of insertion attempts i.e., number of skin punctures needed to successfully insert a peripheral intravenous catheter
Patient's satisfaction | The time frame for the outcome measure patient´s satisfaction for each participant is estimated 1 hour in the pre-implementation stage and 1 hour in the post-implementation stage.
  Arbitrary Likert scale 0-5
Patient's experience of pain | The time frame for the outcome measure patient´s experience of pain for each participant is estimated 1 hour in the pre-implementation stage and 1 hour in the post-implementation stage.
  Numerical Rating Scale (NRS) scale 0-10
Durability | The time frame for the outcome measure durability for each participant is estimated 4 hours in the pre-implementation stage and 4 hours in the post-implementation stage.
  Is the chemotherpy session completed successfully (yes/no). Defined as intravenous chemotherapy successfully infused with only one peripheral intravenous catheter used.
Intravenous complications | The time frame for the outcome measure intravenous complications for each participant is estimated 4 hours in the pre-implementation stage and 4 hours in the post-implementation stage.
  Intravenous complications such as e.g., infiltration, extravasation, vessel occlusion etc.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juhl-Olsen, MD, PhD, Principal Investigator — Aarhus University Hospital; August Gabriel Wang, MD, DMSc, Principal Investigator — University of the Faroe Islands; Lisa Maria Anderssen, RN, MHS, Principal Investigator — Department of Research, the National Hospital of the Faroe Islands

IPD SHARING:
Plan to Share IPD: No
IPD data can be shared on a collaborative basis, provided the appropriate approvals